CLINICAL TRIAL: NCT02346955
Title: A Phase 1, Open-Label, Multicenter, Multi-Dose Escalation Study of CM-24 (MK-6018) as Monotherapy and In Combination With Pembrolizumab (MK-3475) in Subjects With Selected Advanced or Recurrent Malignancies
Brief Title: Study of CM-24 (MK-6018) Alone and In Combination With Pembrolizumab (MK-3475) in Participants With Selected Advanced or Recurrent Malignancies (MK-6018-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Famewave Ltd. (Industry)
Responsible Party: Sponsor
Organization: KitovPharma (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6018-001; CB-24-01 (Registry Identifier: prior cCAM Biotherapeutics Ltd Protocol Number); MK-6018-001 (Other: Merck Registration Number)
Record Dates: First submitted 2014-12-09; First posted 2015-01-27 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Non-small Cell Lung Carcinoma (NSCLC); Melanoma; Bladder Cancer; Colorectal Cancer; Gastric Cancer; Ovarian Cancer
Keywords: Cancer; Oncology; cCAM Biotherapeutics Ltd; Immunomodulatory therapy; CM-24; Carcinoembryonic Antigen-related Cell Adhesion Molecule 1 (CEACAM1); NSCLC (adenocarcinoma); Uveal; Acral; Mucosal; Cutaneous; Colorectal; Gastric; Ovarian; Bladder; MK-6018-001
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Urinary Bladder Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Neoplasms; Adenocarcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Cohort A Monotherapy Dose Escalation (Experimental): Participants will be enrolled in a staggered manner starting at a dose of 0.01 mg/kg of CM-24 (MK-6018) and continuing to 0.03, 0.1, 0.3, 1.0, 3.0, and 10 mg/kg to determine the recommended Phase 2 dose (RP2D). The dose will be escalated after a 6- to 8-week DLT window. Participants will be treated for 12 weeks during Cycle 1. Afterwards participants with clinical benefit and no dose-limiting toxicites (DLTs) are treated for up to 6 cycles.
  Interventions: Biological: CM-24 (MK-6018)
- Cohort B Combination Dose Escalation (Experimental): Participants will be enrolled at the recommended phase 2 dose (RP2D) of CM-24 (MK-6018), determined by escalation studies, minus 1 dose level of MK-6018 in combination with a fixed dose of 200 mg pembrolizumab. Participants will be escalated to the RP2D of MK-6018 + 200 mg pembrolizumab. If the RP2D of MK-6018 + 200 mg pembrolizumab is not tolerated, the dose of MK-6018 will be de-escalated but will not fall below 1 mg/kg. Participants will be treated for 6 weeks during Cycle 1 and 2. Afterwards participants with clinical benefit and no DLTs are treated for up to 35 cycles.
  Interventions: Biological: CM-24 (MK-6018); Biological: Pembrolizumab (MK-3475)
- Cohort C Monotherapy Expansion (Experimental): Participants with advanced or recurrent cutaneous melanoma will be enrolled and treated at the recommended phase 2 dose of CM-24 (MK-6018) for up to 17 cycles.
  Interventions: Biological: CM-24 (MK-6018)
- Cohort D Monotherapy Expansion (Experimental): Participants with advanced or recurrent colorectal cancer will be enrolled and treated at the recommended phase 2 dose of CM-24 (MK-6018) for up to 17 cycles.
  Interventions: Biological: CM-24 (MK-6018)
- Cohort E Monotherapy Expansion (Experimental): Participants with advanced or recurrent gastric cancer will be enrolled and treated at the recommended phase 2 dose of CM-24 (MK-6018) for up to 17 cycles.
  Interventions: Biological: CM-24 (MK-6018)
- Cohort C1 Combination Expansion (Experimental): Participants with advanced or recurrent cutaneous melanoma will be enrolled and treated at the recommended phase 2 dose of CM-24+ 200 mg of Pembrolizumab for up to 17 cycles and may continue to receive 200 mg of Pembrolizumab as monotherapy for up to an additional 18 cycles (up to 35 total cycles).
  Interventions: Biological: CM-24 (MK-6018); Biological: Pembrolizumab (MK-3475)
- Cohort D1 Combination Expansion (Experimental): Participants with advanced or recurrent colorectal cancer will be enrolled and treated at the recommended phase 2 dose of CM-24+ 200 mg of Pembrolizumab for up to 17 cycles and may continue to receive 200 mg of Pembrolizumab as monotherapy for up to an additional 18 cycles (up to 35 total cycles).
  Interventions: Biological: CM-24 (MK-6018); Biological: Pembrolizumab (MK-3475)
- Cohort E1 Combination Expansion (Experimental): Participants with advanced or recurrent gastric cancer will be enrolled and treated at the recommended phase 2 dose of CM-24+ 200 mg of Pembrolizumab for up to 17 cycles and may continue to receive 200 mg of Pembrolizumab as monotherapy for up to an additional 18 cycles (up to 35 total cycles).
  Interventions: Biological: CM-24 (MK-6018); Biological: Pembrolizumab (MK-3475)
- Cohort F Combination Expansion (Experimental): Participants with advanced or recurrent non-small cell lung adenocarcinoma will be enrolled and treated at the recommended phase 2 dose of CM-24+ 200 mg of Pembrolizumab for up to 17 cycles and may continue to receive 200 mg of Pembrolizumab as monotherapy for up to an additional 18 cycles (up to 35 total cycles).
  Interventions: Biological: CM-24 (MK-6018); Biological: Pembrolizumab (MK-3475)

INTERVENTIONS:
Biological: CM-24 (MK-6018) — humanized IgG4 (kappa) isotype monoclonal antibody against CEACAM1 by intravenous (IV) infusion
  Other Names: Anti-CEACAM1
Biological: Pembrolizumab (MK-3475) — 200 mg of Pembrolizumab by IV infusion
  Other Names: KEYTRUDA®
  Arms: Cohort B Combination Dose Escalation; Cohort C1 Combination Expansion; Cohort D1 Combination Expansion; Cohort E1 Combination Expansion; Cohort F Combination Expansion

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of humanized IgG4 (kappa) isotype monoclonal antibody against CEACAM1 (CM-24 [MK-6018]), administered intravenously as monotherapy and in combination with Pembrolizumab (MK-3475), in participants with selected advanced or recurrent malignancies. Escalating multiple doses will be evaluated to determine the recommended dose for Phase 2 clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥18 years of age
* Participants in the Dose Escalation portion must have one of the following advanced or recurrent malignancies: gastrointestinal (colorectal or gastric); ovarian; melanoma; non-small cell lung adenocarcinoma; or bladder.
* Participants in the Monotherapy Expansion Cohort must have one of the following advanced or recurrent malignancies: cutaneous melanoma showing primary progression following treatment with an anti-programmed cell death (PD) or anti-PDL1 regimen; or anti-PD1 or anti-PD-L1 treatment-naïve colorectal or gastric cancer, including gastroesophageal junction cancer of Siewert Type II and Type III.
* Participants in the Combination Expansion Cohorts must have one of the following advanced or recurrent malignancies: non-small cell lung adenocarcinoma or cutaneous melanoma showing primary progression following treatment with an anti-PD1 or anti-PD-L1 regimen; or anti-PD1 or anti-PD-L1 treatment-naïve colorectal or gastric cancer, including gastroesophageal junction cancer of Siewert Type II and Type III.
* Melanoma with BRAF V600E or V600K mutation-positive melanoma must have progressed on, or were intolerant to, prior BRAF- or MEK-inhibitor therapy
* Must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 with progressing or new tumors since last antitumor therapy
* Must have adequate hematologic, renal, and liver function
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Females must not be pregnant (negative human chorionic gonadotropin test within 72 hours prior to receiving the first dose of study medication) or breastfeeding
* Women of childbearing potential and male participants must agree to use adequate contraception throughout the study and for up to 180 days after study treatment
* An estimated life expectancy of at least 3 months
* Must consent to provide an archival tumor biopsy sample at any time point from screening to study exit
* Must consent to allow the acquisition of new tissue biopsy samples during the study

Exclusion Criteria:

* History of severe hypersensitivity reactions or immune related adverse events to other monoclonal antibodies
* History of other active malignancy within the prior 2 years
* History of insulin-dependent or uncontrolled Diabetes Mellitus
* History of inflammatory bowel disease
* Autoimmune disorders
* Known HIV and/or Hepatitis B or C infections
* Known systemic bleeding or platelet disorder
* Receipt of live vaccines with 4 weeks (28 days) of study
* History or evidence of non-infectious pneumonitis that required steroids or current pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-02; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | From time of first dose until the end of follow-up (up to 123 weeks)
Number of participants discontinuing study drug due to AEs | From time of first dose until the end of follow-up (up to 105 weeks)
Number of participants with a Dose Limiting Toxicity (DLT) | From time of first dose until the end of follow-up (up to 12 weeks)

SECONDARY OUTCOMES:
Maximum drug concentration in serum/plasma (Cmax) | For Cycles 1-35: all infusions at pre-infusion. For Cycle 1 first & fourth infusion: at end of infusion; 1, 4, 8 hours post-infusion; and Days 2, 3, 5, 8 post-infusion. For Cycle 1 fourth infusion also at Days 15, 22, 36 post-infusion.
Time to reach Cmax in serum/plasma (Tmax) | For Cycles 1-35: all infusions at pre-infusion. For Cycle 1 first & fourth infusion: at end of infusion; 1, 4, 8 hours post-infusion; and Days 2, 3, 5, 8 post-infusion. For Cycle 1 fourth infusion also at Days 15, 22, 36 post-infusion.
Terminal-phase elimination half-life in serum/plasma (t1/2) | For Cycles 1-35: all infusions at pre-infusion. For Cycle 1 first & fourth infusion: at end of infusion; 1, 4, 8 hours post-infusion; and Days 2, 3, 5, 8 post-infusion. For Cycle 1 fourth infusion also at Days 15, 22, 36 post-infusion.
Area under the plasma/serum concentration versus time curve from time zero to the last measured time (AUC 0-T) | For Cycles 1-35: all infusions at pre-infusion. For Cycle 1 first & fourth infusion: at end of infusion; 1, 4, 8 hours post-infusion; and Days 2, 3, 5, 8 post-infusion. For Cycle 1 fourth infusion also at Days 15, 22, 36 post-infusion.
Area under the plasma/serum concentration versus time curve from time zero to infinity (AUC 0-∞) | For Cycles 1-35: all infusions at pre-infusion. For Cycle 1 first & fourth infusion: at end of infusion; 1, 4, 8 hours post-infusion; and Days 2, 3, 5, 8 post-infusion. For Cycle 1 fourth infusion also at Days 15, 22, 36 post-infusion.
Objective Response Rate (ORR) defined using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria | From time of screening until the end of follow-up (up to 123 weeks)
Time from ORR to disease progression or death (DOR) | From time of screening until the end of follow-up (up to 123 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (3):
- United States (2):
  - Call for Information (Investigational Site 0003), Los Angeles, California
  - Call for Information (Investigational Site 0004), New Haven, Connecticut
- Merck Sharp & Dohme Co. Ltd., Hod HaSharon, Israel